CLINICAL TRIAL: NCT04482595
Title: A Phase 2 Study of BIO 300 Oral Suspension in Discharged COVID-19 Patients
Brief Title: BIO 300 Oral Suspension in Previously Hospitalized Long COVID Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Humanetics Corporation (Industry)
Collaborators: NYU Langone Health (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL0105-01; 272201800011C-P00005-9999-1 (NIH)
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Long COVID; Pulmonary Fibrosis; Post-acute Respiratory Complications of COVID-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIO 300 Oral Suspension (genistein 1500 mg) (Experimental): BIO 300 Oral Suspension (genistein 1500 mg) will be self-administered daily for 7 days each week for 12 weeks.
  Interventions: Drug: BIO 300 Oral Suspension
- Placebo (Placebo Comparator): BIO 300 Oral Suspension matched placebo will be self-administered daily for 7 days each week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIO 300 Oral Suspension — Suspension of genistein nanoparticles
  Arms: BIO 300 Oral Suspension (genistein 1500 mg)
Drug: Placebo — Matched placebo for BIO 300 Oral Suspension
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, two-arm study to evaluate the safety and efficacy of BIO 300 Oral Suspension (BIO 300) as a therapy to improve lung function in patients that were hospitalized for severe COVID-19-related illness and continue to experience post-acute respiratory complications associated with Long-COVID after discharge. Patients will be randomized 1:1 to receive BIO 300 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Patients hospitalized for COVID-19-related complications ready to be discharged and those within 365 days of discharge (even if the patient was referred to subacute or acute respiratory rehabilitation after discharge)
3. Radiographic signs of lung injury after standard treatment of COVID-19 such as, ground glass opacity, consolidation, or fibrotic shadows at screening
4. Able to perform a PFT and have a DLCO <70% of predicted at screening
5. Able to perform a 6-minute walk test
6. Blood routine, liver and kidney function test values are within the controllable range

   1. Adequate hepatic function as evidenced by ALT, AST and LDH < 2X ULN and bilirubin < 1.5X ULN for the reference lab
   2. Adequate renal function as evidenced by a serum creatinine ≤ 1.5 X ULN for the reference laboratory OR a calculated creatinine clearance of ≥ 60 mL/min by the Cockcroft-Gault Equation
   3. Adequate hematopoietic function as evidenced by white blood cells ≥ 3x10^9 / L and platelets ≥ 100x10^9 / L
7. Female patients of childbearing potential must have a negative pregnancy test at screening
8. Female patients of childbearing potential and male participants with female sexual partners of childbearing potential must agree to use an effective method of non-estrogen-based contraception (e.g., condom and a diaphragm, condom and intrauterine device, condom and Depo-Provera, condom and Nexplanon, or condom and progesterone mini-pill) during the 12-week portion of the study that they are receiving study medication and for 30 days following the last dose of study medication, or to abstain from sexual intercourse during these time periods. Women who have been off estrogen contraceptives for a minimum of 5 days prior to the first scheduled day of study intervention dosing are eligible. A woman not of childbearing potential is one who has undergone bilateral oophorectomies or who is post-menopausal, defined as no menstrual periods for 12 consecutive months
9. Ability of the patient or the patient's legal representative to read and provide written informed consent

Exclusion Criteria:

1. Severe background disease like severe cardiac or pulmonary insufficiency (WHO grade III or IV), severe liver and kidney diseases, severe COPD, severe neurological disease, or concurrent malignancy (other than non-melanoma skin cancer) which is uncontrolled or actively being treated
2. Severe asthma on chronic therapy with biologics or steroids.
3. Prior malignancy in which any thoracic radiotherapy was administered except for partial or tangent breast irradiation for early-stage (stages I or II) breast cancer
4. D-dimer levels of >2,000 ng/mL at screening
5. Use of anti-pulmonary fibrosis drugs (e.g., imatinib, nintedanib, pirfenidone, penicillamine, colchicine, tumor necrosis factor alpha blocker) within 5 days of the first scheduled day of study intervention dosing
6. Use of anti-cytokine release syndrome drugs (e.g., anakinra, sarilumab, siltuximab, tocilizumab and/or lenzilumab) within 5 days of the first scheduled day of study intervention dosing
7. Use of systemic corticosteroids (e.g., prednisone, dexamethasone) within 5 days of the first scheduled day of study intervention dosing
8. An active infection or infection with a fever ≥ 38.5°C within 3 days of the first scheduled day of study intervention dosing
9. Poorly controlled intercurrent illnesses, such as interstitial lung disease, uncontrolled hypertension; poorly controlled diabetes mellitus; unstable angina, myocardial infarction, acute coronary syndrome or cerebrovascular event within 6 months of Screening; history of congestive heart failure (NYHA Class III or IV); severe valvular heart disease; or poorly controlled cardiac arrhythmias not responding to medical therapy or a pacemaker
10. QTc with Fridericia's correction that is unmeasurable, or ≥480 msec on screening ECG. The average QTc from the screening ECG (completed in triplicate) must be <480 msec for the patient to be eligible for the study
11. Patients taking any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes (www.crediblemeds.org) are not eligible if QTc ≥460 msec
12. Patients who have undergone thoracotomy within 4 weeks of Day 1 of protocol therapy
13. Patients that have a known allergy to any of the placebo components
14. Psychiatric conditions, social situations or substance abuse that precludes the ability of the study participant to cooperate with the requirements of the trial and protocol therapy
15. Pregnancy or currently on estrogen-based contraceptives
16. Women who are breastfeeding
17. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in DLCO | 12 Weeks
  Diffusing capacity of the lungs for carbon monoxide (DLCO)

SECONDARY OUTCOMES:
Change in 6 Minute Walk Test | 12 Weeks
  6 minute walk test (6MWT)
Change in FVC | 12 Weeks, 6 Months and 12 Months
  Forced vital capacity (FVC)
Change in St. George's Respiratory Questionnaire (SGRQ) Scores | 12 Weeks, 6 Months and 12 Months
  Patient reported outcome to measure impact on overall health, daily life, and perceived well-being in patients with impaired pulmonary function. Scores range from 0-100 with higher scores indicating more limitations.
Change in Pulmonary Fibrosis on HRCT Scan | 12 Weeks, 6 Months and 12 Months
  Evidence of pulmonary fibrosis on high resolution computerized tomography (HRCT) scans of the lungs based on a 4-point Likert scale, where 0 is no evidence of fibrosis and 3 is severe fibrosis
Incidence of Re-Hospitalization | 12 Months
  Incidence of hospitalization after initial discharge and initiating treatment
All-Cause Mortality | 12 Months
  Mortality at 12 months after initiating treatment
Change in FEV1 | 12 Weeks, 6 Months and 12 Months
  Forced expiratory volume in one second (FEV1)
Change in FEV1/FVC Ratio | 12 Weeks, 6 Months and 12 Months
  Ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC)
Change in 6 Minute Walk Test | 6 Months and 12 Months
  6 minute walk test (6MWT)
Change in Pulse Oximetry at Rest and During the 6MWT | 12 Weeks, 6 Months and 12 Months
  Oxygen saturation (pulse oximetry) at rest and during the 6 minute walk test (6MWT)
Change in DLCO | 6 Months and 12 Months
  Diffusing capacity of the lungs for carbon monoxide (DLCO)
Adverse Events Related to BIO 300 Oral Suspension | 12 Months
  Evaluate the safety of BIO 300 Oral Suspension treatment
Change in Clinical Laboratory Values | 4 Weeks, 8 Weeks, 12 Weeks, 6 Months and 12 Months
  Monitoring of blood serum levels for bilirubin, C-reactive protein (CRP), creatinine, blood urea nitrogen (BUN), cholesterol and triglycerides (all reported as mg/dL)
Change in Clinical Laboratory Values | 4 Weeks, 8 Weeks, 12 Weeks, 6 Months and 12 Months
  Monitoring of blood serum levels for troponin T, d-dimer and ferritin (all reported as ng/mL)
Change in Clinical Laboratory Values for Albumin | 4 Weeks, 8 Weeks, 12 Weeks, 6 Months and 12 Months
  Monitoring of blood serum levels for albumin (g/dL)
Change in Clinical Laboratory Values for Serum Enzymes | 4 Weeks, 8 Weeks, 12 Weeks, 6 Months and 12 Months
  Monitoring of blood serum levels for alkaline phosphatase (ALP), alanine transaminase (ALT), aspartate aminotransferase (AST) and lactate dehydrogenase (LDH) (all reported as Units/L)
Change in Complete Blood Counts with Differential | 4 Weeks, 8 Weeks, 12 Weeks, 6 Months and 12 Months
  Monitoring of white blood cell, red blood cell and platelet counts

OTHER OUTCOMES:
Change in Supplemental Oxygen Use | 12 Weeks, 6 Months and 12 Months
  Prescribed supplemental oxygen flow rate at night, rest and exertion
Change in Duration of Supplemental Oxygen Use | 12 Weeks, 6 Months and 12 Months
  Duration of supplemental oxygen use
Change in Serum Cytokine Expression | 4 Weeks, 8 Weeks, 12 Weeks, 6 Months and 12 Months
  Expression levels of serum-derived cytokines (IL-1b, IL-6, IL-8, TNFa, and TGFb1)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - NYU Langone Health, New York, New York
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No